CLINICAL TRIAL: NCT04367103
Title: Norepinephrine or Phenylephrine for Hypotension in Non-elective Cesarean Section
Brief Title: Norepinephrine for Hypotension in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ShA
Record Dates: First submitted 2020-03-26; First posted 2020-04-29 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Hypotension; Cesarean Section
Keywords: post spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEP group (Active Comparator): Norepinephrine infusion of 0.025 µg/kg/min and 6 µg bolus will be used if BP is reduced 20 % below baseline.
  Interventions: Drug: Norepinephrine
- PHE group (Placebo Comparator): Phenylephrine will be started at 25µg/min immediately after the intrathecal local anaesthetic injection and titrated according to blood pressure and pulse rate.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — prophylaxis for hypotension
  Other Names: noradrenaline
  Arms: NEP group
Drug: Phenylephrine — standerd prophylaxis for hypotension
  Other Names: phenylephrine hydrochloride
  Arms: PHE group

SUMMARY:
Hypotension is a very common consequence of the sympathetic vasomotor block caused by spinal anesthesia for cesarean section. Maternal symptoms such as nausea, vomiting and dyspnea frequently accompany severe hypotension, and adverse effects on the fetus, including depressed APGAR scores and umbilical acidosis, have been correlated with severity and duration of hypotension. Because hypotension is frequent, vasopressors should be used routinely and preferably prophylactically.

DETAILED DESCRIPTION:
Phenylephrine has a potent direct α effect, with virtually no β effects at clinical doses, however when given at higher than required doses, it may induce baroreceptor-mediated bradycardia with a consequent reduction in maternal cardiac output. Although α agonist drugs are the most appropriate agents to treat or prevent hypotension following spinal anaesthesia, those with a small amount of β agonist activity may have the best profile (noradrenaline (norepinephrine) and metaraminol. Phenylephrine is currently recommended due to the amount of supporting data.Noradrenaline is the primary catecholamine released by postganglionic adrenergic nerves. It is a potent α adrenergic agonist, with comparatively modest β agonist activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fall in category 2 and 3 according to the classification of Caesarean section made by Royal College of Obstetrician and Gynaecologists.

Exclusion Criteria:

* Patient refusal either to study enrollment or to spinal anesthesia.

  * Any absolute contraindication to spinal anesthesia e.g. coagulopathy, skin infection at site of injection.
  * Allergy to any of study drugs.
  * Patients with cardiac morbidities, hypertensive disorders or peripartum bleeding
  * BMI > 40 kg/m²
  * Baseline systolic blood pressure < 100 mmHg.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotensive episodes. | 15-20 minutes
  Hypotension is defined as <80% of baseline or systolic blood pressure (SBP) <100 mmHg.

SECONDARY OUTCOMES:
Incidence of maternal bradycardia. | 15-20 minutes
  Bradycardia is defined as heart rate (HR) < 50 beats/min
Incidence of reactive hypertension | 20 minutes
  defined as >120% of baseline.
nausea and vomiting | 20 minutes
  Incidence of nausea and vomiting attacks.
Total dose of vasopressor | 20 minutes
  Total dose of vasopressor used.

OTHER OUTCOMES:
Fetal outcome | at 1, 5 and 8 minutes
  APGAR score
mixed blood gas | 1 minute after delivery
  Umbilical artery and vein blood gas
Admission to neonatal ICU (NICU) | first 24 hours after delivery
  the need for NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Abdellatif, M.D., Study Director — Assiut University; Shimaa A. Husien, M.D., Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt